CLINICAL TRIAL: NCT06464445
Title: Defining Parameters to Optimize Neurostimulation for the Treatment of Pediatric Depression
Brief Title: Optimization of ITBS for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-François Lepage, Full professor, Department of Pediatrics, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-5470
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-08

CONDITIONS: Neuromodulation
Keywords: TMS; repetitive TMS; intermittent Theta Burst Stimulation; Plasticity

STUDY DESIGN:
Intervention Model Description: Repeated Measure Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intermittent theta burst stimulation (iTBS) (Experimental): All participants will understand 3 different iTBS protocols, each separated by one week. The order of the iTBS protocols will be randomized.
  Interventions: Device: Monophasic iTBS; Device: Biphasic iTBS; Device: Monophasic-Long iTBS

INTERVENTIONS:
Device: Monophasic iTBS — iTBS protocol with monophasic-shaped pulses. iTBS parameters:
  * Intensity: 80% of resting motor threshold (rMT)
  * Frequency: 50 Hz
  * Duration of pulse train: 2 seconds
  * Interval between pulse trains: 8 seconds
Device: Biphasic iTBS — iTBS protocol with biphasic-shaped pulses. iTBS parameters:
  * Intensity: 80% of rMT
  * Frequency: 50 Hz
  * Duration of pulse train: 2 seconds
  * Interval between pulse trains: 8 seconds
Device: Monophasic-Long iTBS — iTBS protocol with long monophasic-shaped pulses. iTBS parameters:
  * Intensity: 80% of rMT
  * Frequency: 50 Hz
  * Duration of pulse train: 2 seconds
  * Interval between pulse trains: 8 seconds

SUMMARY:
Repetitive TMS (rTMS) is a well-established method for modulating brain activity. Through successive stimulations in the form of magnetic fields, it is possible to modify the sensitivity of neurons in the brain, also known as cortical excitability. Cortical excitability is important for the induction of brain plasticity, the ability of the brain to reorganize itself and form new connections in response to stimuli. A particular class of rTMS, intermittent theta burst TMS (iTBS), is commonly used to modulate cortical excitability and induce plasticity for therapeutic purposes, notably for treatment-resistant depression.

Different iTBS stimulation parameters can be used to induce plasticity. This study will focus on two parameters, namely, the form and duration of the electromagnetic stimulation. The shape of the electromagnetic pulse refers to how the electromagnetic wave is configured over time, while the duration is simply the period during which this electromagnetic pulse remains active. These parameters are expected to influence the effectiveness of iTBS in modulating cortical activity but remain little studied.

The main aim of this study will be to compare the effectiveness of different stimulation parameters in the induction of plasticity, which will then make it possible to improve the rTMS protocols used for treatment-resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 35 years old
* Be of right manual dominance
* In good health

Exclusion Criteria:

* Have an implant or pacemaker,
* Having tinnitus,
* Have a history of fainting,
* Have already had an epileptic seizure or have a family history of epilepsy,
* Have a known neurological disease,
* Be under psychotropic medication,
* Have suffered from substance abuse or dependence in the last 6 months,
* Have a neurostimulator,
* Have a splinter or metallic implant in the head or the rest of the body,
* Have a cochlear implant,
* Have an automated injection system implanted (insulin pump),
* Have a transdermal patch,
* Have tattoos in the area to be studied,
* Be pregnant or breastfeeding,

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
TMS derived measure of cortical plasticity | Pre-iTBS, Every 5 minutes post iTBS intervention up to 60 minutes post intervention.
  Change in Peak-to-peak motor evoked potential (MEP) amplitude induced by the administration of the test stimulus (stimulation intensity required to produce an MEP of 1 millivolt, approximately 120% of rMT) after iTBS

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche du Centre hospitalier universitaire de Sherbrook, Sherbrooke, Quebec, Canada